CLINICAL TRIAL: NCT00270439
Title: Omentectomy for Treatment of Diabetes Mellitus Type 2
Brief Title: Omentectomy for the Treatment of Diabetes Mellitus Type 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: United States Surgical Corporation (Other)
Responsible Party: Dr. William Richards, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050967
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus Type 2; Dyslipidemia; Hypercholesterolemia; Obesity
Keywords: Obesity; Omentectomy; Diabetes Mellitus Type 2; Laparoscopic; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias; Hypercholesterolemia; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): Removed omentum of patients with type 2 diabetes
  Interventions: Procedure: removal of omentum

INTERVENTIONS:
Procedure: removal of omentum — patients with type 2 diabetes had their omentum removed
  Other Names: laparoscopic omentum removal

SUMMARY:
The purpose of this study is to determine whether laparoscopic removal of the omentum (thin layer of fat inside the abdomen) will significantly improve insulin resistance in patients with non-insulin dependent type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Clinical studies have shown that central obesity is one of the strongest associations with Type II diabetes. Measurement of waist circumference at Vanderbilt was one of the most effective clinical measures of presence of type II diabetes and response to gastric bypass in a recent study. This central obesity points to the omentum as one of the major culprits for development and perpetuation of type II diabetes in humans. [1]

Animal studies at Vanderbilt have shown in normal size dogs that surgical removal of the visceral fat (Omentectomy):

* Decreases basal hepatic glucose production by nearly 40%
* Results in decreased FFA delivery to the liver
* Increases glucose utilization by peripheral insulin dependent tissues, predominantly skeletal muscle. [2] The animal studies were started to pursue the positive results seen by Swedish investigators who randomized 50 patients to either gastric banding or to gastric banding with omentectomy. At 2 years both groups had statistically similar weight loss but the patients in the omentectomy group had 2 to 3 times the improvements in oral glucose tolerance, insulin sensitivity and fasting plasma glucose as compared to control subjects. [3] They concluded that omentectomy, when combined with gastric banding in morbidly obese patients had a significant positive effects on the glucose and insulin metabolism.

Why does the removal of visceral fat (a very small percentage of the animal's weight) cause a 40% increase in peripheral glucose metabolism? The omentum is known to be a repository for macrophages and the increase in macrophage numbers is proportional to the increase in adiposity in humans. Both macrophages and adipocytes produce adipokines and cytokines that are known to influence glucose and insulin metabolism. The omentum is also known to be the major contributor of Free Fatty Acids into the portal circulation which adversely affects the hepatic insulin resistance.

Resection of the visceral fat which holds more numbers of the macrophages which in turn release the cytokines that preferentially disturb glucose metabolism should in theory then result in a marked improvement in glucose and fat metabolism.

Hypothesis Removal of visceral fat (omentectomy) will significantly improve type II Diabetes and dyslipidemia.

Specific Aim 1: Determine the improvement in glucose metabolism in patients with type II diabetes using Minimal model study at baseline and at 3 months post surgery Specific Aim 2: Determine the improvement in control of type II diabetes by measuring HgbA1c levels and the amount of oral medications taken to control their diabetes 3, 6 and 12 months post surgery.

Specific aim 3: Determine the improvement in lipids by measuring fasting serum total cholesterol, HDL, LDL and Triglycerides at 0, 3, 6, and 12 months post surgery.

Specific Aim 4: Determine the effect of omentectomy on markers of inflammation (C- reactive protein, interleukin 6) at 3, 6, and 12 months post op. These labs will be drawn but not assayed until we see the effects on insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55
* BMI 30-50
* Dyslipidemia
* Non-insulin dependent Type 2 diabetes Mellitus on oral hypoglycemics only

Exclusion Criteria:

* Medicare patients
* significant hepatic enzyme elevations (more than 50% of upper limits of normal)
* serum creatinine >1.5 mg/dl
* history of ketoacidosis or current metabolic acidosis
* current use of oral anticoagulants
* positive pregnancy test (β-human chorionic gonadotrophin) for females
* intercurrent infections
* taking drugs that are known to affect carbohydrate or lipid metabolism (e.g. steroids, high dose Niacin, β-adrenergic receptor agonists, but does not include anti-diabetic drugs)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity as measured by the minimal model and HOMA score | one year post procedure

SECONDARY OUTCOMES:
Improvement in dyslipidemia | One year post procedure
Decreased use of oral hypoglycemics | One year post procedure

CONTACTS AND LOCATIONS:
Overall Officials: William O Richards, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Thorne A, Lonnqvist F, Apelman J, Hellers G, Arner P. A pilot study of long-term effects of a novel obesity treatment: omentectomy in connection with adjustable gastric banding. Int J Obes Relat Metab Disord. 2002 Feb;26(2):193-9. doi: 10.1038/sj.ijo.0801871. PMID 11850750
- [Background] Torquati A, Lutfi R, Abumrad N, Richards WO. Is Roux-en-Y gastric bypass surgery the most effective treatment for type 2 diabetes mellitus in morbidly obese patients? J Gastrointest Surg. 2005 Nov;9(8):1112-6; discussion 1117-8. doi: 10.1016/j.gassur.2005.07.016. PMID 16269382
- [Background] Hansen, E., et al., Omentectomy Improves Insulin Sensitivity in Skeletal Muscle in vivo. 2005, Abstract Society of University Surgeons.
- [Background] Bergman RN, Finegood DT, Ader M. Assessment of insulin sensitivity in vivo. Endocr Rev. 1985 Winter;6(1):45-86. doi: 10.1210/edrv-6-1-45. No abstract available. PMID 3884329
- [Background] Bonora E, Kiechl S, Willeit J, Oberhollenzer F, Egger G, Targher G, Alberiche M, Bonadonna RC, Muggeo M. Prevalence of insulin resistance in metabolic disorders: the Bruneck Study. Diabetes. 1998 Oct;47(10):1643-9. doi: 10.2337/diabetes.47.10.1643. PMID 9753305
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Derived] Fabbrini E, Tamboli RA, Magkos F, Marks-Shulman PA, Eckhauser AW, Richards WO, Klein S, Abumrad NN. Surgical removal of omental fat does not improve insulin sensitivity and cardiovascular risk factors in obese adults. Gastroenterology. 2010 Aug;139(2):448-55. doi: 10.1053/j.gastro.2010.04.056. Epub 2010 May 7. PMID 20457158